Retrospective, Multicenter, Observational Study to

Evaluate Current Treatment patterns and Outcomes in

Japanese Patients with Locally Advanced or Metastatic

Urothelial Carcinoma Treated with First-line Avelumab

Maintenance

| rincipal Inve | stigator |
|---------------|----------|
| PPD | |
| PPD | |

Statistical Analysis Plan (SAP)

Version: 1.1

Date: 21-Dec-2022

| Research Sponsor Medical Affairs, Oncology, Pfizer Japan Inc. | Approval date : |
|---|---|
| Chief statistical analyst CR Data Science Department, Clinical Research Center, Real World Evidence Business Headquarters, EPS Co., Ltd. | Approval date: |

# Table of Contents

| 1 | PU | RPOSE | 3 |
|---|---|---|---|
| 2 | An | alysis Environment | 3 |
| 2 | .1 | Statistical analysis, tabulation software | 3 |
| 3 | Ove | erview of Study Design | 3 |
| 3 | .1 | Primary objectives | 3 |
| 3 | .2 | Secondary objectives | 3 |
| 3 | .3 | Study design | 3 |
| C | CI | | 4 |
| 4 | En | lpoints | 4 |
| 4 | .1 | Primary endpoint | 4 |
| 4 | .2 | Secondary endpoints | 4 |
| 5 | Ha | ndling of study population and data | 5 |
| 5 | .1 | Analysis set/populations | 5 |
| 5 | .2 | Handling of missing values | 5 |
| 5 | .3 | Handling of data on the number of days | 5 |
| 5 | .4 | Steroid equivalent dose (prednisolone-equivalent dose) | 5 |
| 5 | .5 | Derived variable | 6 |
| 5 | .6 | Variable conversion | 13 |
| 6 | Sta | tistical processing | 13 |
| 6 | .1 | Confidence interval/significance level | 13 |
| 6 | .2 | Multiple comparisons/multiplicity | 13 |
| 6 | .3 | Details of statistical analysis | |
| 6 | .3.1 | Summary statistics | 13 |
| 6 | .3.2 | Number of digits | 13 |
| 7 | Ana | alysis of primary endpoints | |
| 8 | | tistical Analysis of Secondary endpoints | |
| 8 | .1 | Efficacy endpoints | |
| 8 | 1.1 | Time to treatment failure (TTF) of avelumab | |
| | 1.2 | Real-world progression-free survival (rwPFS) | |
| | .1.3 | Objective Response Rate (ORR) | |
| | .1.4 | Real-world progression-free survival from chemotherapy (rwPFS-c) | |
| | .2 | Safety endpoints | |
| | .2.1 | Corticosteroid therapy for immune-related adverse events (irAEs) | |
| | .2.2 | Premedication for potential infusion-related reaction of avelumab | |
| | .2.3 | Treatment for infusion-related reaction of avelumab | |

| 8. | 2.4 | Regimen after avelumab maintenance therapy | 24 |
|---|---|---|---|
| 8. | 2.5 | Hematological test (from the start of the first anticancer chemotherapy) | 25 |
| CCI | | | 26 |
| | | | 29 |
| 10 | 0.1 | Cause of death | 29 |
| 11 | Ref | erences | 30 |
| | | vision record | 30 |

#### 1 PURPOSE

The purpose of this statistical analysis plan is to define the details of statistical methods for the statistical analysis activities related to "Retrospective, Multicenter, Observational Study to Evaluate Current Treatment patterns and Outcomes in Japanese Patients with Locally Advanced or Metastatic Urothelial Carcinoma Treated with First-line Avelumab Maintenance - (Protocol No.: B9991048)" (hereinafter referred to as "Study").

# 2 Analysis Environment

# 2.1 Statistical analysis, tabulation software

The software and version expected to be used are shown below. The software and version eventually used should be clearly stated in the analysis results.

| Items | Software and Version |
|----------------------|----------------------|
| OS | Microsoft Windows 10 |
| Statistical analysis | SAS Ver. 9.4 |
| software | |
| Tabulation software | Microsoft Excel 365 |

# 3 Overview of Study Design

#### 3.1 Primary objectives

To describe the demographic and baseline disease characteristics of patients with locally advanced or metastatic UC treated with avelumab as 1L maintenance therapy in a real-world clinical setting.

#### 3.2 Secondary objectives

- 1) To evaluate the effectiveness of 1L avelumab maintenance therapy for patients with locally advanced or metastatic UC treated in Japan.
- 2) To describe clinical usage of corticosteroid for immune-related adverse events (irAEs) observed during avelumab therapy and after the last administration of avelumab therapy.
- 3) To describe premedication and treatment for infusion-related reaction of avelumab.
- 4) To describe the patterns of subsequent UC therapy.

# 3.3 Study design

This study is a multicenter, non-interventional, retrospective, medical chart review of

locally advanced or metastatic UC patients who were prescribed avelumab as 1L maintenance therapy between 24 February 2021 and 30 November 2021 in Japan. All decisions regarding clinical management and treatment of the participating patients were made by the investigator as part of standard care in a real-world clinical setting and were not contingent upon the patient's participation in the study. Data will be collected if available per study site.

- Index date: The date of first prescription for avelumab between 24 February 2021
   (launch date of avelumab) and 30 November 2021
- Observation period: Patients will be followed from index date to 30 Jun 2022



#### 4 Endpoints

#### 4.1 Primary endpoint

 Patient characteristics at baseline (at the initiation of first line chemotherapy and the initiation of avelumab maintenance therapy)

#### 4.2 Secondary endpoints

#### Efficacy endpoints

- Time to treatment failure (TTF) of avelumab
- · Real-world progression-free survival (rwPFS)
- Objective Response Rate (ORR)
- · Real-world progression-free survival from chemotherapy (rwPFS-c)

## Safety endpoints

- Corticosteroid therapy for immune-related adverse events (irAEs)
- Premedication for potential infusion-related reaction of avelumab
- Treatment for infusion-related reaction of avelumab
- Regimen after avelumab maintenance therapy
- Hematological test (At the start of first-line chemotherapy/ immediately before the first

avelumab administration/ at the start of fourth cycle of avelumab treatment/ at the time of PD judgment (at the latest test during the observation period for those continuing avelumab treatment without disease progression)

# 5 Handling of study population and data

#### 5.1 Analysis set/populations

Among patients who were enrolled in the study and received maintenance avelumab treatment between 24 February 2021 and 30 November 2021, patients meeting all the inclusion criteria will be analyzed.

#### 5.2 Handling of missing values

An absence of data for analysis will be treated as missing values, and no special imputation processing will be performed using statistical methods.

However, if there are specifications for handling of missing values in subsequent each specification, they are followed.

#### 5.3 Handling of data on the number of days

The number of days from the start date to the target date will be calculated as follows:

- The target date is earlier than the start date = Target date Start date
- The target date is on or after the start date = Target date Start date + 1

If the data for "year" and "month" among the date data are missing, no calculation will be performed.

If the data on "day" of the date is missing, data will be substituted by 1.

The number of days in one month is converted to 30.

#### 5.4 Steroid equivalent dose (prednisolone-equivalent dose)

The corticosteroid-equivalent dose (prednisolone-equivalent) is calculated as the dose of the starting drug × prednisolone conversion ratio, according to the table below.

| General name | Corresponding dose | Prednisolone |
|--------------------|--------------------|------------------|
| | (mg) | conversion ratio |
| Cortisone | 25 | 0.2 |
| Hydrocortisone | 20 | 0.25 |
| Prednisolone | 5 | 1 |
| Methylprednisolone | 4 | 1.25 |
| Triamcinolone | 4 | 1.25 |

| Dexamethasone | Approximately 0.75 | 6.67 |
|---------------|--------------------|------|
| Betamethasone | Approximately 0.75 | 6.67 |

# 5.5 Derived variable

The items and definitions of variables whose derivation is necessary at the time of statistical analysis are shown below.

# Continuous variable

| Item | Derivation method |
|---|---|
| from the end date of first-line | Start date of initial administration with avelumab – end date of first-line chemotherapy administration + 1 |
| chemotherapy (days) | End date of first-line chemotherapy administration — start date of first-line chemotherapy administration + 1 |
| treatment) of corticosteroid (days) | End date of corticosteroid administration — start date of corticosteroid administration + 1 |
| avelumab (TTF) | Defined as the period from the date of start of avelumab to the date of end of treatment* for any reasons including death. If there is no record of end of treatment, patients will be censored at the date of last observation during the study period. *The following sensitivity analysis will also be performed. Considering its clinical meaning, "interruption due to being well-controlled" does not correspond to "treatment failure"; it should be treated as an event on the day when the death or discontinuation was observed prior to the last observation date. If no death or discontinuation occurred before the date of the last observation, data will be censored at the date of the last observation. |
| | Defined as the period from the start date of<br>avelumab maintenance therapy to the date of first |

| | , |
|---|---|
| | disease progression (clinical evaluation based on imaging examinations, laboratory tests, and pathological tests, as well as other evaluations by the investigators of each institution) or death from any cause, whichever occurs earlier. If there is no record of death or disease progression, patients on second or later lines (following avelumab maintenance therapy) will be censored at the start of the second-line treatment, and patients on only avelumab maintenance therapy will censored at the date of the last visit during the |
| | study, based on the medical record. |
| Real-world progression-free survival from chemotherapy (rwPFS-c) | Defined as the period from the start date of first- line chemotherapy to the date of first disease progression (clinical evaluation based on imaging examinations, laboratory tests, and pathological test, as well as other evaluations by the investigators of each institution) or death from any cause, whichever occurs earlier. If there is no record of death or disease progression, patients on second or later lines (following avelumab maintenance therapy) will be censored at the start of the second-line treatment, and patients on only avelumab maintenance therapy will censored at the date of the last visit during the study, based on the medical record. |
| Starting dose of corticosteroid | Calculate according to "5.4 Steroid equivalent dose |
| (Steroid equivalent dose) | (prednisolone-equivalent dose." |
| Duration of treatment of | |
| corticosteroid (days) | administration of the first steroid drug + 1 |
| Duration of treatment of avelumab maintenance (days) | Last administration date – date of first administration + 1. |
| Duration of treatment of each regimen (days) | Last administration date – date of first administration + 1. |

# Categorical variable

| Item | Derivation method |
|---|---|
| Age (2 divisions) | Age is divided into the following categories: |
| | <65 years/65 years or older |
| Site of primary tumor (2 | The primary site is divided into the following |
| divisions) | categories: |
| | "upper urinary tract" for renal pelvis or ureter |
| | "lower urinary tract" for bladder and urethra |
| Tumor histological type (2) | The histological types are divided into the following |
| | categories. |
| | "Urothelial carcinoma" for urothelial carcinoma |
| | "Non-urothelial carcinoma" for adenocarcinoma, |
| | squamous cell carcinoma, small cell carcinoma, or |
| | others |
| Presence or absence of visceral | "Presence" will be selected if the metastatic site is |
| metastasis | "lung," "liver," "adrenal gland," "pancreas," "kidney," |
| | "spleen," or "other" which is regarded as visceral |
| | metastasis. If the metastatic site is not regarded as |
| | visceral metastasis, "absence" will be selected. |
| Presence or absence of non- | " Presence" will be selected if the metastatic site is |
| visceral metastasis | "bone," "distant lymph nodes," or "other" which is |
| | regarded as non-visceral metastasis. If the |
| | metastatic site is not regarded as non-visceral |
| | metastasis, "absence" will be selected. |
| ECOG Performance Status at | ECOG Performance Status at start of first-line |
| start of first-line | chemotherapy is categorized as follows. |
| chemotherapy (1) | 0/1 or higher |
| *For at the start of avelumab | |
| administration, " at the start | |
| of first-line chemotherapy | |
| administration" should be read | |
| as "at the start of avelumab | |
| administration." | |
| Performance Status at start of | ECOG Performance Status at start of first-line |
| first-line chemotherapy (2) | chemotherapy is categorized as follows. |
| *For at the start of avelumab | 0/1/2 or higher |

| administration, " at the start | | | | |
|---|---|---|---|---|
| of first-line chemotherapy | | | | |
| administration" should be read | | | | |
| as "at the start of avelumab | | | | |
| administration." | | | | |
| Number of cycles in first-line | Number of cy | vcles in first-li | ine chemother | apy is |
| chemotherapy (3 divisions) | divided into | the following | categories. | |
| | 3 or less/4 to | _ | S | |
| Karnofsky performance status | Karnofsky pe | erformance st | atus is divided | l into the |
| (2 divisions) | following c | | | |
| (2 divisions) | | | | |
| D 1 1 | <80%/>=80% | | | C 11 |
| Bajorin risk classification | | | is categorized | as follows |
| | | number of ris | sk factors. | |
| | <risk factors<="" td=""><td></td><td></td><td></td></risk> | | | |
| | · Visceral m | etastasis is "p | resent" | |
| | <ul> <li>Karnofsky</li> </ul> | performance | status is "<80 | %" |
| | If there is no | risk factor, "( | ) (no risk facto | or)". |
| | If there is on | e risk factor, ' | '1 (single risk | factor)". |
| | If there are t | wo risk factor | rs, "2 (two risk | factors)". |
| Clinical stage classification: | Clinical stage is categorized using primary tumor (T | | | |
| Bladder | factor), regin | al lymph nod | es (N factor), d | listant |
| | metastasis (I | M factor) as fo | ollows. | |
| | Primary | Reginal | Distant | Clinical |
| | tumor (T | lymph | metastasis | stage |
| | factor) | nodes (N | (M factor) | |
| | Ta | factor)<br>N0 | M0 | 00 |
| | Tis | N0<br>N0 | M0 | 0a<br>0is |
| | T1 | N0 | MO | I |
| | T2a, T2b | N0 | M0 | II |
| | T3a, T3b, | N0 | MO | IIIA |
| | T4a | 271 | Mo | TTT A |
| | T1, T2a,<br>T2b, T3a, | N1 | M0 | IIIA |
| | T3b, T4a | | | |
| | T1, T2a, | N2, N3 | M0 | IIIB |
| | T2b, T3a, | | | |
| | T3b, T4a | A . NT | Mo | TX7A |
| | T4b<br>Any T | Any N<br>Any N | M0<br>M1a | IVA<br>IVA |
| | Any T | Any N<br>Any N | M1b | IVB |
| | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | 1 1111 / 1 1 | 11110 | 1110 |

| Urethra | factor), reginal lymph nodes (N factor), distant | | | |
|---|---|---|---|---|
| | metastasis (M factor) as follows. | | | |
| | Primary<br>tumor (T<br>factor) | Reginal<br>lymph<br>nodes (N | Distant<br>metastasis<br>(M factor) | Clinical stage |
| | | factor) | | |
| | Ta | N0 | M0 | 0a |
| | Tis | NO | M0 | 0is |
| | T1<br>T2 | N0<br>N1 | M0<br>M0 | I |
| | T1, T2 | N1 | MO | III |
| | T3 | N0, N1 | MO | III |
| | T4 | N0, N1 | MO | IV |
| | Any T | N2 | MO | IV |
| | Any T | Any N | M1 | IV |
| Clinical stage classification: | Clinical stag | e is categoriz | ed using prima | ary tumor (T |
| Renal pelvis, Ureter | factor), reginal lymph nodes (N factor), distant | | | |
| | metastasis (M factor) as follows. | | | |
| | Primary | Reginal | Distant | Clinical |
| | tumor (T | lymph | metastasis | stage |
| | factor) | nodes (N<br>factor) | (M factor) | |
| | Ta | N0 | MO | 0a |
| | Tis | N0 | MO | 0is |
| | T1 | N0 | MO | Ι |
| | T2 | N0 | M0 | II |
| | Т3 | N0 | M0 | III |
| | T4 | N0 | M0 | IV |
| | Any T | N1, N2 | M0 | IV |
| | Any T | Any N | M1 | IV |
| Treatment-free interval: Time | Time from th | ne end date of | first-line chen | notherapy to |
| from the end date of first-line | the start dat | e of avelumal | administratio | on is divided |
| chemotherapy to the start date | into the follo | wing categori | es. | |
| of avelumab administration (3 | <4 weeks/4 to 10 weeks/>10 weeks | | | |
| divisions) | | | | |
| Response (avelumab | Determination of the best overall response to | | | |
| maintenance) | avelumab maintenance is categorized as following: | | | |
| | "Objective response" when "CR" or "PR." | | | |
| | "Non-objective response" when "SD" of "PD" | | | |
| Response (first-line | | | overall respons | |
| chemotherapy) | chemotherapy is categorized as following: | | | g: |

| | "Objective response" when "CR" or "PR." |
|---|---|
| | "Non-objective response" when "SD" of "PD" |
| Best overall response to first- | Determination of the best overall response to first- |
| line chemotherapy (2) | line chemotherapy is categorized as following: |
| | CR+PR/SD |
| Presence or absence of | "Presence" will be selected when "prednisolone" is |
| prednisolone | selected for the corticosteroid administration drug |
| | name, and "absence" will be selected when "No" is |
| | selected for the drug name. |
| Presence or absence of | "Presence" will be selected when |
| methylprednisolone | "methylprednisolone" is selected for the |
| | corticosteroid administration drug name, and |
| | "absence" will be selected when "No" is selected for |
| | the drug name. |
| Presence or absence of | "Presence" will be selected when "betamethasone" is |
| betamethasone | selected for the corticosteroid administration drug |
| | name, and "absence" will be selected when "No" is |
| | selected for the drug name. |
| Presence or absence of | "Presence" will be selected when "dexamethasone" is |
| dexamethasone | selected for the corticosteroid administration drug |
| | name, and "absence" will be selected when "No" is |
| | selected for the drug name. |
| Presence or absence of | "Presence" will be selected when "hydrocortisone" is |
| hydrocortisone | selected for the corticosteroid administration drug |
| | name, and "absence" will be selected when "No" is |
| | selected for the drug name. |
| Presence or absence of others | "Presence" will be selected when "other" is selected |
| | for the corticosteroid administration drug name, and |
| | "absence" will be selected when "No" is selected for |
| | the drug name. |
| Presence or absence of | "Absence" will be selected if the prednisolone- |
| treatment with non-high-dose | equivalent starting dose is 40 mg or higher. |
| corticosteroid | "Presence" will be selected if it is less than 40 mg. |
| Presence or absence of | "Absence" will be selected if the prednisolone- |
| treatment with high-dose | equivalent starting dose is less than 40 mg. |
| corticosteroid | "Presence" will be selected if it is 40 mg or higher. |

| Presence or absence of steroid | "Absence" will be selected if the prednisolone- |
|---|---|
| pulse therapy | equivalent starting dose is less than 625 mg. |
| | "Presence" will be selected if it is 625 mg or higher. |
| NLR | Neutrophil count (/μL)/lymphocyte count (/μL) |
| Hematological test (Red blood | Hematological test (Red blood cell count, hemoglobin, |
| cell count, hemoglobin, | hematocrit, white blood cell count, neutrophil count, |
| hematocrit, white blood cell | eosinophil, basophil, monocyte, lymphocyte count, |
| count, neutrophil count, | platelet count, CRP, total protein, albumin, AST, |
| eosinophil, basophil, monocyte, | ALT, LDH, BUN, creatinine, Na, K, Cl, NLR) is |
| lymphocyte, platelet count, | categorized as following: |
| CRP, total protein, albumin, | < median/≥ median |
| AST, ALT, LDH, BUN, | |
| creatinine, Na, K, Cl, NLR (2 | |
| divisions) | |
| Hemoglobin (g/dL) (2) | Hemoglobin is divided into the following categories: |
| | <10 g/dL/>=10 g/dL |
| White blood cell count (2) | White blood cell count is divided into the following |
| | categories: |
| | <8000/μL/>=8000/μL |
| NLR (2) | NLR is divided into the following categories: |
| | <3/>=3 |
| NLR (3) | NLR at the start of the first-line chemotherapy and |
| | at the start of first cycle of avelumab is divided into |
| | the following categories, regarding NLR at the start |
| | of first cycle of avelumab as a starting point. |
| | "Low→Low" when changed from NLR <3 (Low) to |
| | NLR <3 (Low), |
| | "Low→High" when changed from NLR <3 (Low) to |
| | NLR ≥3 (High), |
| | "High→Low" when changed from NLR ≥3 (High) to |
| | NLR <3 (Low), |
| | "High→High" when changed from NLR ≥3 (High) to |
| | NLR ≥3 (High) |

#### 5.6 Variable conversion

No variable conversion is performed.

# 6 Statistical processing

# 6.1 Confidence interval/significance level

The significance level of hypothesis testing will be two-sided 5%. A two-sided 95% confidence interval will be calculated if interval estimation is performed.

#### 6.2 Multiple comparisons/multiplicity

Multiplicity will not be adjusted.

#### 6.3 Details of statistical analysis

# 6.3.1 Summary statistics

If summary statistics is described in this plan, the following values will be calculated unless otherwise specified.

Number of subjects, number of subjects with missing, mean, standard deviation, minimum value, quartile point (25% point, 50% point [median], 75% point), maximum value

#### 6.3.2 Number of digits

Percentages will be rounded to 1 decimal place for the fraction distribution, unless the details of the individual items are specified. Among the summary statistics (number of subjects, mean standard deviation, minimum value, quartiles (25% point, 50% point [median], 75% point), and maximum value), the mean, standard deviation, and quartiles (25% point, 50% point [median], 75% point) are rounded up to where a decimal place is one digit below the original data.

# 7 Analysis of primary endpoints

# 7.1 Patient characteristics at baseline (at the start of the first-line chemotherapy and at the start of the avelumab administration)

Target: Analysis set

populatio

n

Endpoints : 1) Primary lesion at initial diagnosis

# Categorical Variable

Site of the primary tumor

Histology of primary lesion<sup>1)</sup>

Presence or absence of variant histology

Subtype

Histologic dysplasia

Two-step grade

Three-step grade

Histological depth

Presence/absence of definitive treatment of primary lesion

Treatment

Surgery

# 2) At the start of the first-line chemotherapy

# Continuous variable

Number of cycles of first-line chemotherapy

Number of cycles at the evaluation of best overall response to firstline chemotherapies

Treatment-free interval: Time from the end of first-line chemotherapy to the start date of avelumab administration (days)

Duration of first-line chemotherapy (days)

# Categorical Variable

**ECOG Performance Status** 

Karnofsky performance status (%)

Karnofsky performance status (2 divisions)

Bajorin risk classification

Staging (TNM classification)

Primary tumor (T factor)

Metastases to regional lymph nodes (N factor)

Distant metastasis (M factor)

Clinical Stage

Bladder

Urethra

Renal pelvis and ureter

Presence/absence of distant metastasis

distant metastasis site

Presence or absence of visceral metastasis

Presence or absence of non-visceral metastasis

Number of metastatic organs

Number of metastases in one organ

Number of distant metastases

Presence/absence of local recurrence

Regimen for first-line chemotherapy

Best overall response to first-line chemotherapies

#### 3) At the start of avelumab administration

#### Continuous variable

Age

# Categorical Variable

Gender

**ECOG Performance Status** 

Karnofsky performance status (%)

Karnofsky performance status (2 divisions)

Bajorin risk classification

Staging (TNM classification)

Primary tumor (T factor)

Metastases to regional lymph nodes (N factor)

Distant metastasis (M factor)

Clinical Stage

Bladder

Urethra

Renal pelvis and ureter

Presence/absence of distant metastasis

Site of distant metastasis

Presence or absence of visceral metastasis

Presence or absence of non-visceral metastasis

Presence or absence of past medical history<sup>2)</sup>

Details of past medical history

Details of past medical history of auto-immune disease

Details of other medical history

Presence or absence of complication<sup>2)</sup>

**Details of Complication** 

Details of complication of auto-immune disease

Details of other complications

Presence/absence of concomitant medication with steroid or immunosuppressant

Details of concomitant drugs using steroids and immunosuppressants

1) If multiple selections are made, the following will be used to determine the tissue type:

Small cell carcinoma > Urothelial carcinoma > It is determined by the order of predominant histological type in terms of quantity.

- If there is any "small cell carcinoma," "small cell carcinoma" is adopted. (If both small cell carcinoma and urothelial carcinoma are selected, small cell carcinoma is adopted.)
- ii. If there is no "small cell carcinoma," and "urothelial carcinoma" exists, "urothelial carcinoma" is adopted.
- iii. If neither "small cell carcinoma" nor "urothelial carcinoma" exists, the tissue type listed in the EDC comment section as the predominant tissue type in terms of quantity is adopted.
- 2) If disease is cured by the start of avelumab administration, it is regarded as past medical history. If it is continued after the administration of avelumab, it is regarded as complication.

Statistical

The following tabulation will be performed for end points.

analysis

Summary statistics will be calculated for continuous variables.

A frequency table (number of subjects, proportion (%)) will be prepared for categorical variables.

A frequency table (number of subjects and proportion (%)) will be prepared also for the details of past medical history of auto-immune disease, other past medical history, complication of auto-immune disease, other complication, and concomitant medications of steroids and immunosuppressants.

# [Division of categorical variables]

| Factor | Division |
|---------|----------|
| 1 40001 | Biviolon |

| Site of the primary tumor | bladder/urethra/renal pelvis/ureter |
|---|---|
| Histology of primary lesion | Urothelial carcinoma/adenocarcinoma/squamous |
| | cell carcinoma/small cell carcinoma/other |
| Presence or absence of variant | presence/absence/unknown |
| histology | |
| Subtype | nested, including large |
| | nested/microcystic/micropapillary/lymphoepithel |
| | ioma-like/plasmacytoid/signet ring |
| | cell/diffuse/sarcomatoid/giant cell/poorly |
| | differentiated/lipid-rich/clear cell/other |
| Histologic dysplasia | two step grades (low grade, high grade)/three step |
| | grades (G1, G2, G3)/unknown |
| Histologic dysplasia: two-step grade | low grade/high grade |
| Histologic dysplasia: three-step | G1/G2/G3 |
| grade | |
| Histological depth | Bladder: |
| | pTX/pT0/pTa/pTis/pT1/pT2a/pT2b/pT3a/pT3bpT |
| | 4a/pT4b |
| | Urethra: pTX/pT0/pTa/pTis/pT1/pT2/pT3/pT4 |
| | Renal pelvis: |
| | pTX/pT0/pTa/pTis/pT1/pT2/pT3/pT4 |
| | Ureter: pTX/pT0/pTa/pTis/pT1/pT2/pT3/pT4 |
| Presence/absence of definitive | absence/presence/unknown |
| treatment of primary lesion | |
| Treatment | surgery/others |
| Surgery | Data will be aggregated based on the combination |
| | of the data obtained. |
| Gender | male/female |
| ECOG Performance Status | 0/1/2/3/4 |
| Karnofsky performance status (%) | 100/90/80/70/60/50/40/30/20/10/0 |
| Karnofsky performance status (2 | <80%/>=80% |
| divisions) | |
| Bajorin risk classification | 0 (no risk factor)/1 (single risk factor)/2 (two risk |
| | factors) |
| Staging (TNM classification): | Bladder: |
| Primary tumor (T factor) | T0/Ta/Tis/T1/T2a/T2b/T3a/T3b/T4a/T4b/unknow |

| | n/other |
|---|---|
| | Urethra: T0/Ta/Tis/T1/T2/T3/T4/ unknown/other |
| | Renal pelvis: T0/Ta/Tis/T1/T2/T3/T4/ |
| | unknown/other |
| | Ureter: T0/Ta/Tis/T1/T2/T3/T4/unknown/other |
| Staging (TNM classification): | Bladder: N0/N1/N2/N3/unknown |
| | Urethra: NO/N1/N2/unknown |
| Metastases to regional lymph nodes (N factor) | |
| (N factor) | Renal pelvis: N0/N1/N2/unknown |
| C. (TDVD 1 | Ureter: N0/N1/N2/unknown |
| Staging (TNM classification): | Bladder: M0/M1a/M1b/unknown/other |
| Distant metastasis (M factor) | Urethra: M0/M1/unknown/other |
| | Renal pelvis: M0/M1/unknown/other |
| | Ureter: M0/M1/unknown/other |
| Clinical Stage: Bladder | 0a/0is/I/II/IIIA/IIIB/IVA/IVB |
| Clinical Stage: Urethra | 0a/0is/I/II/III/IV |
| Clinical Stage: Renal pelvis | 0a/0is/I/II/III/IV |
| Clinical Stage: Ureter | 0a/0is/I/II/III/IV |
| Presence/absence of distant | presence/absence/unknown |
| metastasis | |
| Site of distant metastasis | lung/liver/adrenal/pancreas/kidney/spleen/bone/ |
| | distant lymph nodes/other |
| Presence or absence of visceral | presence/absence |
| metastasis | |
| Presence or absence of non-visceral | presence/absence |
| metastasis | |
| Number of metastatic organs | Single organ metastasis/multiple organ |
| | metastasis |
| Number of metastases in one organ | single/multiple |
| Number of distant metastases | single ("single organ metastasis" and |
| | "single")/multiple ("multiple organ metastasis" + |
| | "single organ metastasis" and "multiple") |
| Presence/absence of local recurrence | presence/absence/unknown |
| Presence or absence of past medical | presence/absence/unknown |
| history | |
| Details of past medical history | interstitial lung disease/chronic obstructive |
| | pulmonary disease (COPD)/auto-immune |

| | disease/cerebrovascular disorder/cardiovascular |
|---|---|
| | disorder/diabetes mellitus/other |
| Presence or absence of complication | presence/absence/unknown |
| Details of Complication | interstitial lung disease/chronic obstructive |
| | pulmonary disease (COPD)/auto-immune |
| | disease/cerebrovascular disorder/cardiovascular |
| | disorder/diabetes mellitus/other |
| Presence/absence of concomitant | presence/absence/unknown |
| medication with steroid or | |
| immunosuppressant | |
| Regimen for first-line chemotherapy | gemcitabine + cisplatin/gemcitabine + |
| | carboplatin/MVAC/dose dense-MVAC/other |
| Best overall response to first-line | CR/PR/SD/PD |
| chemotherapies | |

# 8 Statistical Analysis of Secondary endpoints

# 8.1 Efficacy endpoints

## 8.1.1 Time to treatment failure (TTF) of avelumab

Target: Analysis set

populatio

n

Endpoint : Time to treatment failure (TTF) of avelumab

Statistical : For the endpoint, the median and its 95% confidence interval will be

analysis calculated using the Kaplan–Meier method. In addition, the Kaplan–

Meier curve will be plotted, and the TTF rate for every 2 months and its 95% confidence interval will be calculated. Greenwood's formula

will be used to calculate the confidence interval for the TTF rate.

In order to evaluate the overall observation period of the study, the

median observation period will be calculated by estimating the reverse KM curve in which censoring patients are regarded as

patients with events and patients with events are regarded as

censoring patients.

In addition, as a sensitivity analysis, "interruption due to being well-controlled" will be treated as an event based on the day when death or discontinuation was observed before the date of the last observation, and if no death or discontinuation or death occurred before the date of the last observation, data will be censored at the date of the last observation.

#### 8.1.2 Real-world progression-free survival (rwPFS)

Target : Analysis set

populatio

n

Endpoint : Real-world progression-free survival (rwPFS)

Statistical : For the endpoint, the median and its 95% confidence interval will be analysis calculated using the Kaplan–Meier method. In addition, the Kaplan–

Meier curve will be plotted, and the rwPFS rate for every 2 months and its 95% confidence interval will be calculated. Greenwood's formula will be used to calculate the confidence interval for the

rwPFS rate.

In order to evaluate the overall observation period of the study, the median observation period will be calculated by estimating the reverse KM curve in which censoring patients are regarded as patients with events and patients with events are regarded as censoring patients.

#### 8.1.3 Objective Response Rate (ORR)

Target: Analysis set

populatio

n

Endpoint : Objective Response Rate (ORR)

Statistical : For the end point in the avelumab maintenance and first-line

analysis chemotherapy, the number of patients included, the number of

responders, and the response rate will be calculated along with its 95% confidence interval. In addition, summary statistics will be calculated for the number of cycles at the time of determination of

best overall response.

The denominator for each proportion (%) will be the analysis set, and patients with missing value for the end point will be excluded from

the denominator.

Clopper-Pearson method will be used to calculate the confidence

#### interval.

#### [Division of categorical variables]

| Factor | 区分 |
|----------|--------------------------------------------|
| Response | Objective response/ Non-objective response |

# 8.1.4 Real-world progression-free survival from chemotherapy (rwPFS-c)

Target: Analysis set

populatio

n

Endpoint

Real-world progression-free survival from chemotherapy (rwPFS-c)

Statistical analysis

For the endpoint, the median and its 95% confidence interval will be calculated using the Kaplan–Meier method. In addition, the Kaplan–Meier curve will be plotted, and the rwPFS-c rate for every 2 months and its 95% confidence interval will be calculated. Greenwood's formula will be used to calculate the confidence interval for the

In order to evaluate the overall observation period of the study, the median observation period will be calculated by estimating the reverse KM curve in which censoring patients are regarded as patients with events and patients with events are regarded as censoring patients.

#### 8.2 Safety endpoints

#### 8.2.1 Corticosteroid therapy for immune-related adverse events (irAEs)

rwPFS-c rate.

Target : Analysis set

populatio

n

Endpoint : <u>Continuous variable</u>

Corticosteroid starting dose<sup>1)</sup> (prednisolone equivalent)

Duration of treatment with corticosteroid (days)

Categorical variable

Presence/absence of corticosteroid administration to irAE

Presence or absence of prednisolone

Presence or absence of methylprednisolone

Presence or absence of betamethasone
Presence or absence of dexamethasone
Presence or absence of hydrocortisone
Presence or absence of others
Details of other drugs

Presence or absence of treatment with non-high-dose corticosteroid (prednisolone-equivalent starting dose is less than 40)

Presence or absence of treatment with high-dose corticosteroid (prednisolone-equivalent starting dose is 40 mg or higher)

Presence or absence of steroid pulse therapy (prednisolone-equivalent starting dose is 625 mg or higher)

1) As the Instruction on the EDC and the EDC operation manual describes the instruction to "enter starting dose (dose change after the start of tapering is unnecessary)", it is likely that only the starting dose is collected. However, if there is any entry of dose change (dose increase) according to the instruction, the dose should be used to determine the starting dose of corticosteroid (the maximum value of the starting dose of each case (including administration change) is used as the starting dose of corticosteroid. When administrations of multiple drugs overlap with the duration of administration, the total dose is considered to be the value of the starting dose.

Statistical analysis

The following aggregation will be performed for endpoints:
Summary statistics will be calculated for continuous variables.

A frequency table (number of cases, proportion [%]) will be created for categorical variables.

A frequency table (number of cases, proportion (%)) will also be created for details regarding other drugs.

# [Category Variable Classification]

| Factor | Division |
|-------------------------------------|----------------------------------|
| Presence/absence of corticosteroid | Absence/Presence/Unknown/Missing |
| administration to irAE | |
| Presence or absence of prednisolone | Absence/Presence |
| Presence or absence of | Absence/Presence |
| methylprednisolone | |

| Presence or absence of | Absence/Presence |
|--------------------------------------|------------------|
| betamethasone | |
| Presence or absence of | Absence/Presence |
| dexamethasone | |
| Presence or absence of | Absence/Presence |
| hydrocortisone | |
| Presence or absence of others | Absence/Presence |
| Presence or absence of treatment | Presence |
| with non-high-dose corticosteroid | |
| Presence or absence of treatment | Presence |
| with high-dose corticosteroid | |
| Presence or absence of steroid pulse | Presence |
| therapy | |

# 8.2.2 Premedication for potential infusion-related reaction of avelumab

Target : Analysis set

populatio

n

Endpoint : Premedication for potential infusion-related reaction of avelumab

Detailed name of the drug

Detailed name of the other drug

Statistical : A frequency table (number of cases, proportion (%)) will be created

analysis for the endpoints.

# [Division of categorical variables]

| Factor | Division |
|------------------------------|----------------------------------------------|
| Presence or absence of | Absence/Presence/Unknown |
| premedication for potential | |
| infusion-related reaction of | |
| avelumab | |
| Detailed name of the drug | Acetaminophen/diphenhydramine |
| | hydrochloride/chlorpheniramine maleate/Other |

#### 8.2.3 Treatment for infusion-related reaction of avelumab

Target : Analysis set

populatio

n

Endpoint : Treatment for infusion-related reaction of avelumab

Detailed name of the drug

Statistical : A frequency table (number of cases, proportion (%)) will be created

analysis for the endpoints.

#### [Division of categorical variables]

| Factor | Division |
|----------------------------------|--------------------------|
| Presence or absence of treatment | Absence/Presence/Unknown |
| for infusion-related reaction of | |
| avelumab | |

## 8.2.4 Regimen after avelumab maintenance therapy

Target: Analysis set

populatio

n

Endpoint : <u>Continuous variable</u>

Duration of Treatment after avelumab maintenance therapy (Days)

Categorical variable

Presence/absence of UC treatment after avelumab maintenance therapy

Regimen after avelumab maintenance therapy

Statistical : The following aggregation will be performed for the end point.

analysis For continuous variables, summary statistics will be calculated for

each treatment. A frequency table (number of subjects, proportion (%)) will be created for the presence or absence of UC treatment after

avelumab maintenance therapy.

A frequency table (number and proportion (%)) will be created for the second-line, third-line and subsequent treatment regimens for the second-line and subsequent treatment after avelumab maintenance

therapy.

In addition, a listing of patients will be prepared.

# [Division of categorical variables]

| Factor | Division |
|----------------------------------|----------------------------------|
| Presence or absence of treatment | Absence/Presence/Unknown/Missing |
| after avelumab maintenance | |
| therapy | |

#### 8.2.5 Hematological test (from the start of the first anticancer chemotherapy)

Target : Analysis set

populatio

n

Endpoint : red blood cell count ( $\times 10^4/\mu L$ )

hemoglobin (g/dL)

hematocrit (%)

white blood cell count (/µL)

neutrophil count (/µL)

eosinophil (%)

basophil (%)

monocyte (%)

lymphocyte count (/µL)

platelet count ( $\times 10^4/\mu L$ )

CRP (mg/dL)

total protein (g/dL)

albumin (g/dL)

AST (IU/L)

ALT (IU/L)

LDH (U/L)

BUN (mg/dL)

creatinine (mg/dL)

Na (mEq/L)

K (mEq/L)

Cl (mEq/L)

NLR

Statistical analysis

Summary statistics of end points will be calculated by each timing of

evaluation (At the start of first line chemotherapy/ immediately

before the first avelumab administration/ at the start of fourth cycle of avelumab treatment/ at the time of PD judgment (at the latest test

during the observation period for those continuing avelumab

treatment without disease progression).







| <br> |
|------|





Confidential



# 11 References

- Bajorin DF, Dodd PM, Mazumdar M, et al. Long-term survival in metastatic transitional-cell carcinoma and prognostic factors predicting outcome of therapy. J Clin Oncol. 1999 Oct;17(10):3173-81.
- Pre-pembrolizumab neutrophil-to-lymphocyte ratio (NLR) predicts the efficacy of second-line pembrolizumab treatment in urothelial cancer regardless of the prechemo NLR

Cancer Immunol Immunother. 2022 Feb;71(2):461-471. doi: 10.1007/s00262-021-03000-8. Epub 2021 Jul 7.

# 12 Revision record

| Version | Date of creation | Reason for revision |
|---------|------------------|-------------------------------------------------|
| Version | 2 November 2022 | New document |
| 1.0 | EPSCo., Ltd. | |
| | Hanae Uemura | |
| Version | 21 December 2022 | |
| 1.1 | EPSCo., Ltd. | Correction of typographical errors |
| | Hanae Uemura | Addition of determination rules for tumor |
| | | histological type |
| | | Addition of the starting dose of corticosteroid |

End of document